CLINICAL TRIAL: NCT01700985
Title: A Double-Blind, Randomized, Single Center, Vehicle-Controlled, Parallel Group Study to Determine the Efficacy and Safety of 122-0551 in Subjects With Plaque Psoriasis Receiving Two Weeks of Treatment
Brief Title: A Study to Determine the Efficacy and Safety of 122-0551 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122-0551-203
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis; Plaque Psoriasis
Keywords: psoriasis; plaque psoriasis; 122-0551; steroid
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 122-0551 (Experimental)
  Interventions: Drug: 122-0551
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: 122-0551 — Applied twice daily for two weeks
  Arms: 122-0551
Drug: Vehicle — Applied twice daily for two weeks
  Arms: Vehicle

SUMMARY:
Corticosteroids are one of the mainstays of treatment for subjects with corticosteroid-responsive dermatoses such as psoriasis. This study has been designed to determine and compare the efficacy and safety of a formulation of 122-0551 versus the corresponding Vehicle in subjects with stable plaque psoriasis after twice daily dosing for 14 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of stable plaque psoriasis
* Subject has an ODS score for the Treatment Area of 3 or 4 at study start

Exclusion Criteria:

* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
* Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
* Subject has used any phototherapy, photo-chemotherapy or systemic corticosteroid therapy within 30 days prior to study start
* Subject has used any systemic methotrexate, retinoids, cyclosporine or analogous products within 90 days prior to study start
* Subject has used any systemic biologic therapy for the treatment of psoriasis within 5 half-lives of the biologic prior to study start
* Subject had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to study start
* Subject has used topical body (excluding the scalp) psoriasis therapy including coal tar, anthralin, steroids, retinoids, vitamin D analogs (e.g., Dovonex®) within 14 days prior to study start
* Subject has used emollients/moisturizers on areas to be treated within four hours prior to clinical evaluation at study start
* Subject is currently using lithium or Plaquenil (hydroxychloroquine)
* Subject is currently using a beta-blocking medication (e.g., propranolol) or ACE (e.g., lisinopril) inhibitor at a dose that has not been stabilized
* Subject is pregnant, lactating, or is planning to become pregnant during the study
* Subject is currently enrolled in an investigational drug or device study
* Subject has used an investigational drug or investigational device treatment within 30 days prior to study start
* Subject has been previously enrolled in this study and treated with a test article

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syd Dromgoole, PhD, Study Director — Therapeutics, Inc.
Locations (2):
- United States (2):
  - Therapeutics Clinical Research, San Diego, California
  - DermResearch, Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 2012 to September 2012
  The location of clinical sites included dermatology clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Period: Overall Study
Arm/Group | 122-0551 | Vehicle
Started | 23 | 21
Completed | 23 | 20
Not Completed | 0 | 1
Not completed — Incarcerated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analyses are based on the Safety population. All participants enrolled in the study who were dispensed and applied test article at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | 122-0551 | Vehicle | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (14.3) | 48.6 (14.9) | 50.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 19 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 20 | 15 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Disease Severity (ODS) Score
Description: The percentage of subjects with ODS "treatment success" at EOS where EOS is the subject's last completed visit. "Treatment success" is defined as an ODS of 0 or 1. ODS is measured on a 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe/very severe.
Time Frame: baseline and Day 15 (End of Study - EOS)
Population: Analysis shown is the Intent-to-treat (ITT) population, defined as all participants who were randomized, applied at least one dose, and had at least one follow-up visit after the Baseline visit. One study participant (VEH group) did not return to the clinic (incarcerated) following Visit 1 (baseline visit) and was excluded from the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 | Vehicle
Number analyzed (Participants) | 23 | 20
percentage of participants | 52.2 | 0.0
Statistical Analysis 1: Comparison: 122-0551 vs Vehicle; Test type: Superiority; p < 0.0001, Fisher Exact

2. Secondary Outcome: ODS "Treatment Success" at Day 8 and Day 15
Description: The percentage of subjects with ODS "treatment success" at Day 8 and Day 15. "Treatment success" is defined as an ODS of 0 or 1. ODS is measured on a 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe/very severe.
Time Frame: baseline, Day 8, and Day 15
Population: Analysis shown is the Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 | Vehicle
Number analyzed (Participants) | 23 | 20
percentage of participants
  Day 8 | 0.0 | 0.0
  Day 15 | 52.2 | 0.0
Statistical Analysis 1: Comparison: 122-0551 vs Vehicle; Test type: Superiority; p < 0.0001, Fisher Exact — At Day 15

3. Secondary Outcome: ODS "Improved" at Day 8 and Day 15
Description: The percentage of subjects rated "improved" with respect to ODS at Days 8 and 15. "Improved" is defined as at least a 2 grade decrease in ODS score relative to baseline. ODS is measured on a 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe/very severe.
Time Frame: baseline, Day 8, and Day 15
Population: Analysis shown is the Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 | Vehicle
Number analyzed (Participants) | 23 | 20
percentage of participants
  Day 8 | 0.0 | 0.0
  Day 15 | 52.2 | 0.0
Statistical Analysis 1: Comparison: 122-0551 vs Vehicle; Test type: Superiority; p < 0.0001, Fisher Exact — At Day 15

4. Secondary Outcome: "Treatment Success" for Clinical Signs and Symptoms of Psoriasis
Description: The percentage of subjects rated "treatment success" for each of the clinical signs and symptoms of psoriasis (scaling, erythema, plaque elevation) at Days 8 and 15. "Treatment success" is defined as a score of 0 or 1 based on a 5-point ordinal scale where 0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe.
Time Frame: baseline, Day 8 and Day 15
Population: Analysis shown is the Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 | Vehicle
Number analyzed (Participants) | 23 | 20
percentage of participants
  Scaling (Day 8) | 21.7 | 0.0
  Scaling (Day 15) | 60.9 | 0.0
  Erythema (Day 8) | 0.0 | 0.0
  Erythema (Day 15) | 21.7 | 0.0
  Plaque Elevation (Day 8) | 8.7 | 0.0
  Plaque Elevation (Day 15) | 56.5 | 0.0

5. Secondary Outcome: "Improved" for Clinical Signs and Symptoms of Psoriasis
Description: The percentage of subjects rated "improved" for each of the clinical signs and symptoms of psoriasis (scaling, erythema, plaque elevation, pruritus) at Days 8 and 15. "Improved" is defined as at least a 2 grade decrease in score based on a 5-point ordinal scale where 0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe.
Time Frame: baseline, Day 8 and Day 15
Population: Analysis shown is the Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 | Vehicle
Number analyzed (Participants) | 23 | 20
percentage of participants
  Scaling (Day 8) | 26.1 | 0.0
  Scaling (Day 15) | 73.9 | 0.0
  Erythema (Day 8) | 0.0 | 0.0
  Erythema (Day 15) | 34.8 | 0.0
  Plaque Elevation (Day 8) | 4.3 | 0.0
  Plaque Elevation (Day 15) | 56.5 | 0.0

6. Secondary Outcome: Change in % Body Surface Area (BSA) With Psoriasis
Description: Changes in % BSA with active psoriasis in the Treatment Area at Days 8 and 15.
Time Frame: baseline, Day 8 and Day 15
Population: Analysis shown is the Intent-to-treat (ITT) population. The mean percent BSA at baseline was 4.8 for the active group (122-0551) and 4.6 for the vehicle group.
Measure: Mean (Standard Deviation); unit: Change in percent BSA
Arm/Group | 122-0551 | Vehicle
Number analyzed (Participants) | 23 | 20
Change in percent BSA
  Day 8 | -0.3 (0.69) | 0.0 (0.0)
  Day 15 | -1.3 (2.07) | 0.0 (0.32)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from study Day 1 (enrollment/first dose) to study completion (Day 15) or early participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The Safety population included all participants enrolled in the study who were dispensed and applied the test article at least once; all participants enrolled in the study applied the first application in the clinic and were included in the Safety population.
Arm/Group | 122-0551 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 1/23 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 122-0551 (N=23) | Vehicle (N=21)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 30 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.